CLINICAL TRIAL: NCT03910647
Title: the Effect of Daily Use of Proton Pump Inhibitors for One Month on Renal Function
Brief Title: Effect of Daily Use Proton Pump Inhibitors for One Month on Kidney Function
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, hanan monsif israil markous, director .samir kamal abdel-hameed, Assiut University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PPIs with kidney function
Record Dates: First submitted 2019-04-03; First posted 2019-04-10 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Proton Pump Inhibitor Allergy
MeSH Terms: interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pantoprazole with normal kidney function (Experimental): use pantoprazole for one month and after one month i will do for them kidney functions test
  Interventions: Drug: pantoprazole
- pantoprazole with abnormal kidney function (Experimental): use pantoprazole for one month and after one month i will do for them kidney functions test
  Interventions: Drug: pantoprazole

INTERVENTIONS:
Drug: pantoprazole — effect of this drug on renal function
  Other Names: Protonix

SUMMARY:
The aim of this study to: evaluate the association between prolonged use of PPI and adverse renal outcomes on patients with normal renal function and others with abnormal renal function

DETAILED DESCRIPTION:
Proton pump inhibitors (PPIs) are one of the most widely used classes of drugs and are prescribed primarily for gastric acid-related diseases, eradication of Helicobacter pylori, and prevention of nonsteroidal anti-inflammatory drug (NSAID)-induced gastropathy,and gastroesophagial reflux diseases . Although PPIs have an excellent overall safety profile, some severe adverse effects, which include bone fracture, dementia, myocardial infarction, infections, micronutrient deficiencies, and kidney diseases,PPIs may trigger acute interstitial nephritis,a potentially sever adverse event commonly associated with acute kidney injury The increase in prescription and inadequate use of this class of medication calls for studies on the effects of prolonged PPI therapy on renal function.

ELIGIBILITY:
Inclusion Criteria:

* patients with peptic ulcer disease or gastroesophagial reflux with normal l renal function
* patients with peptic ulcer disease or gastroeosophagial reflux with abnormal renal function

Exclusion Criteria:

* 1- cigarette smoker: Cigarette smoking status was defined categorically as current,former, or never smoker at baseline.

  2-biabetic patients: diabetes mellitus is defined by a fasting blood glucose concentration >_ 126 mg/dl ,random glucose level of >200 mg/dl.

  3-patients take corticosteroid 4-patients with hypersensitivity to these drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
kidney function | one month
  eGFR=175xage(y/0)x^(-0.203)xplasma creatinine (mg/dl)x^(-1.154)

CONTACTS AND LOCATIONS:
Overall Officials: samir k abdel-hameed, Study Director — Assiut University; mohammad y kobeisy, prof, Study Director — Assiut University

REFERENCES:
- [Background] Desbuissons G, Deray G, Mercadal L. [Proton pump inhibitors and kidney]. Nephrol Ther. 2018 Apr;14 Suppl 1:S115-S124. doi: 10.1016/j.nephro.2017.06.005. Epub 2017 Dec 20. French. PMID 29274872
- [Background] Mak SK, Loo CK, Wong PN, Lo KY, Tong GM, Lam EK, Wong AK. A retrospective study on efficacy of proton-pump inhibitor-based triple therapy for eradication of Helicobacter pylori in patients with chronic renal failure. Singapore Med J. 2003 Feb;44(2):74-8. PMID 14503780